CLINICAL TRIAL: NCT03306498
Title: Plasma Free Amino Acids in Patients With Hepatic Encephalopathy and Its Impact on Disease Outcomes.
Brief Title: Plasma Free Amino Acids in Patients With Hepatic Encephalopathy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Hamed Goda, Specialist, Assiut University
Other Study IDs: amino acids in liver cirrhosis
Record Dates: First submitted 2017-10-05; First posted 2017-10-11 (Actual); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Hepatic Encephalopathy
Keywords: plasma free amino acids
MeSH Terms: conditions — Hepatic Encephalopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- hepatic encephalopathy patients: The following will be administered to this group of patients rifaximin 550 tablets b.i.d Lactulose syrup 5cm b.i.d Enema b.i.d for 3 days
- hepatic encephalopathy patients-amino: The following will be administered to this group of patients rifaximin 550 tablets b.i.d Lactulose syrup 5cm b.i.d Enema b.i.d plus Aminoleban (8% amino acids infusion) b.i.d for 3 days
  Interventions: Drug: Aminoleban (8% amino acids infusion)

INTERVENTIONS:
Drug: Aminoleban (8% amino acids infusion) — Each 1000ml of AMINOLEBAN contains: Aminoacetic acid - 9.0 g L-alanine -- 7.5 g L-arginine Hydrochloride (HCl) -- 7.3 g (L-arginine equivalent) -- (6.0 g) L-cysteine HCl monohydrate -- 0.4 g (L-cysteine equivalent) -- (0.3 g) L-histidine HCl monohydrate -- 3.2 g (L-histidine equivalent)-- (2.4 g) L-isoleucine -- 9.0 g L-leucine -- 11.0 g L-Lysine HCl -- 7.6 g (L-lysine equivalent) -- (6.1 g) L-methionine -- 1.0 g L-phenylalanine -- 1.0 g L-proline -- 8.0 g L-serine -- 5.0 g L-threonine -- 4.5 g L-tryptophan -- 0.7 g L-valine -- 8.4 g Water for injection q.s -- 1000 m
  Groups: hepatic encephalopathy patients-amino

SUMMARY:
This is study to investigate the plasma free amino acids profile in patients with decompensated liver cirrhosis and hepatic encephalopathy and its relation to the nutritional state of these patients.

* To investigate the plasma free amino acids relation to the nutritional state of patients with liver cirrhosis and hepatic encephalopathy.
* To determine the effectiveness, cost, cost-benefit and in-hospital prognosis of branched chain amino acid (BCAA) infusion as an adjuvant to conventional mainstay therapy in the treatment of hepatic encephalopathy due to liver cirrhosis.
* To determine the effectiveness of branched chain amino acid (BCAA) infusion on improving amino acid imbalance and Fischer ratio (Branched chain amino acids/Aromatic amino acids ratio).

DETAILED DESCRIPTION:
Alterations in amino acid profiles observed in patients with liver cirrhosis are very specific and markedly differ from those observed in other disorders..

Until present time the treatment of hepatic encephalopathy is mainly aimed at reducing the production and intestinal absorption of ammonia by antibiotics and non-absorbable disaccharides, although the available data indicate a low success rate of these strategies.

Beneficial effects of branched chain amino acids supplementation (BCAA) may be more pronounced in patients with marked depression of BCAA and/or low Branched chain amino acids/Aromatic amino acids (BCAA/AAA) ratio in extracellular fluid.

It also may be suggested that the beneficial effect of long term intake of BCAA on hepatic encephalopathy demonstrated in clinical studies is related to improved muscle mass and nutritional status.

The current recommendation only includes oral BCAA to patients with liver disease who are intolerant to standard protein intake.

The rationale for this limitation is based on the fact that in the mentioned randomized trials, hepatic encephalopathy was not part of the inclusion criteria. Additionally, the positive effect was difficult to interpret as it was observed on compound end points, which combine survival, hospitalization, and cirrhosis complications. From these results, it is not possible to ascertain the role of BCAA in hepatic encephalopathy, which patients benefit and to what extent .

For this reason, the investigators designed this study to assess effectiveness of BCAA in improving clinical, nutritional and laboratory status of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient has decompensated liver cirrhosis
* Patient has overt hepatic encephalopathy

Exclusion Criteria:

1. Protein losing enteropathy.
2. Neurological conditions that make the assessment of hepatic encephalopathy difficult

   1. Parkinson's disease
   2. Alzheimer's disease
   3. Concomitant stroke
3. Gastrointestinal Bleeding requiring blood transfusion

   -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients known to be cirrhotic admitted at Al-Rajhi liver hospital at Assiut university by hepatic encephalopathy
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-12-15 (Estimated); Primary Completion 2018-12-15 (Estimated); Study Completion 2019-02-15 (Estimated)

PRIMARY OUTCOMES:
Amino acid profile in hepatic encephalopathy | 24 hours
  Measuring the level of plasma different free amino acids in hepatic encephalopathy patients

SECONDARY OUTCOMES:
Relation between amino acids and nutrition | 24 hours
  Study the relation between amino acid profile and nutritional status of hepatic encephalopathy patients.
IV Amino acids infusion effect | up to 1 week
  Investigating the prognosis and in-hospital mortality of patients with hepatic encephalopathy following the use of IV Amino acids infusion for 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad H Salem, MD, Study Chair — Assiut University; Mahmoud HG Abdel-Rahman, Master, Principal Investigator — Assiut University; Sahar M Hassany, Study Director — Assiut University

REFERENCES:
- [Background] Als-Nielsen B, Gluud LL, Gluud C. Non-absorbable disaccharides for hepatic encephalopathy: systematic review of randomised trials. BMJ. 2004 May 1;328(7447):1046. doi: 10.1136/bmj.38048.506134.EE. Epub 2004 Mar 30. PMID 15054035
- [Background] Als-Nielsen B, Koretz RL, Kjaergard LL, Gluud C. Branched-chain amino acids for hepatic encephalopathy. Cochrane Database Syst Rev. 2003;(2):CD001939. doi: 10.1002/14651858.CD001939. PMID 12804416
- [Background] Charlton M. Branched-chain amino-acid granules: can they improve survival in patients with liver cirrhosis? Nat Clin Pract Gastroenterol Hepatol. 2006 Feb;3(2):72-3. doi: 10.1038/ncpgasthep0392. No abstract available. PMID 16456570
- [Background] Dam G, Ott P, Aagaard NK, Vilstrup H. Branched-chain amino acids and muscle ammonia detoxification in cirrhosis. Metab Brain Dis. 2013 Jun;28(2):217-20. doi: 10.1007/s11011-013-9377-3. Epub 2013 Jan 15. PMID 23315357
- [Background] Holecek M. Ammonia and amino acid profiles in liver cirrhosis: effects of variables leading to hepatic encephalopathy. Nutrition. 2015 Jan;31(1):14-20. doi: 10.1016/j.nut.2014.03.016. Epub 2014 Mar 30. PMID 25220875
- [Background] Phongsamran PV, Kim JW, Cupo Abbott J, Rosenblatt A. Pharmacotherapy for hepatic encephalopathy. Drugs. 2010 Jun 18;70(9):1131-48. doi: 10.2165/10898630-000000000-00000. PMID 20518580
- [Background] Wright G, Jalan R. Management of hepatic encephalopathy in patients with cirrhosis. Best Pract Res Clin Gastroenterol. 2007;21(1):95-110. doi: 10.1016/j.bpg.2006.07.009. PMID 17223499